CLINICAL TRIAL: NCT07117929
Title: Effects of Pulsed Electromagnetic Field Therapy on Meniscal Healing, Symptom Relief, and Knee Function in Patients With Isolated Meniscal Tears: A Randomized Controlled Trial
Brief Title: Effects of Pulsed Electromagnetic Field Therapy on Meniscal Healing, Symptom Relief, and Knee Function
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Patrick Shu-Hang YUNG, Professor and Chairman, Department of Orthopaedics & Traumatology, Faculty of Medicine, The Chinese University of Hong Kong, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024.622-T; 22230771 (Other Grant/Funding Number: Health and Medical Research Fund)
Record Dates: First submitted 2025-07-28; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Meniscal Tears
Keywords: meniscal injuries; meniscus tear; meniscal injury
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PEMF Group (Active Comparator): 1. PEMF Therapy: Participants will undergo active PEMF therapy sessions lasting 10 minutes each, conducted twice weekly for 16 sessions, with a specified PEMF device (QuantumTX Pte Ltd, Singapore).
  2. Exercise Therapy: All participants will be provided with the same standardised home exercise protocol.
  Interventions: Device: Active PEMF; Other: Exercise
- Control Group (Sham Comparator): 1. Sham PEMF Therapy: Participants will undergo sham PEMF therapy sessions lasting 10 minutes each, conducted twice weekly for 16 sessions, with a specified PEMF device (QuantumTX Pte Ltd, Singapore).
  2. Exercise Therapy: All participants will be provided with the same standardised home exercise protocol.
  Interventions: Device: Sham PEMF; Other: Exercise

INTERVENTIONS:
Device: Active PEMF — PEMF: 1.5mT, 10Hz, 10 minutes
  Arms: PEMF Group
Device: Sham PEMF — PEMF 0mT, 0Hz, 10 minutes
  Arms: Control Group
Other: Exercise — Standardised home exercise protocol

SUMMARY:
The goal of this clinical trial is to learn if pulsed electromagnetic field (PEMF) combined with home exercise improves healing and function in adults with meniscus tears. The main questions it aims to answer are:

1. Does PEMF therapy help heal meniscus tears, as seen on MRI scans?
2. Does PEMF therapy subjectively reduce knee pain, improve movement, and enhance quality of life?
3. Does PEMF therapy objectively help patients perform daily activities more easily?

Researchers will compare PEMF therapy against a sham (inactive) treatment to determine if it provides additional benefits.

Participants will:

* Be assigned randomly to either the PEMF group (active treatment) or the sham PEMF group (inactive, but identical in appearance)
* Receive either real PEMF therapy or sham treatment twice a week for 8 weeks (each session lasts 10 minutes).
* Follow a standard home exercise program to strengthen their knees.
* Have their knee function, pain levels, and healing progress checked through MRI scans, questionnaires, imaging and physical tests.
* Return for 3 follow-up visits after the 8-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18-60
* Clinical history, signs, and symptoms indicative of a meniscal tear
* MRI confirmation of a non-displaced, and unilateral meniscal tear
* Meniscal tears located within red-white and white-white zones
* Willingness to adhere to a 8-week regimen of PEMF and exercise therapy
* Ability to provide written informed consent

Exclusion Criteria:

* Congenital discoid meniscus confirmed by MRI
* Complex, oblique, flap, or displaced bucket handle tears confirmed by MRI
* Meniscal root tears confirmed by MRI
* Evidence of partial healing on baseline MRI
* Presence of mechanical symptoms (e.g., locking or catching)
* Acute onset exacerbation of knee symptoms (e.g., severe pain or swelling)
* Surgical intervention during the therapy session
* Knee axis deformities that necessitate surgical correction
* Prior surgery or fracture in the affected limb within the past 12 months
* Severe radiographic knee OA (Kellgren-Lawrence scale ≥2)
* Implanted electronic medical devices (e.g., pacemakers or cochlear implants) • Current pregnancy or intention to become pregnant during the study period

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Between-group difference in mean change of intrameniscal fluid-equivalent signal area at 6 months post-intervention, as assessed by MRI. | Baseline to 6 months post intervention
  A musculoskeletal radiologist, blinded to the participants' group assignments and clinical details, will perform these assessments using fat- suppressed T2-weighted imaging. The primary imaging endpoint will be the between-group difference in the mean change of the intrameniscal fluid-equivalent signal area (mm2) from baseline to 6 months. The fluid-equivalent signal area will be delineated and quantified using standardized region-of-interest (ROI) methods on consecutive slices encompassing the original tear site.

SECONDARY OUTCOMES:
Change in Knee Injury and Osteoarthritis Outcome Score (KOOS) Scores for Pain, Symptoms, Activities of Daily Living, Sport/Recreation Function, and Knee-Related Quality of Life | Baseline to 1-, 2-, 6-, and 12-months post intervention
  The KOOS score is a 42-item patient-reported outcome measure assessing five subscales: Pain (9 items, score range 0-100), Symptoms (7 items, 0-100), Activities of Daily Living (17 items, 0-100), Sport/Recreation Function (5 items, 0-100), and Quality of Life (4 items, 0-100). Each subscale is scored separately from 0 (extreme problems) to 100 (no problems), with higher scores indicating better outcomes.
Change in Western Ontario Meniscal Evaluation Tool (WOMET) Scores for Physical Symptoms, Sports/Work/Lifestyle, and Emotional Domains | Baseline, 1, 2, 6, and 12 months post-intervention
  The WOMET is a 16-item patient-reported questionnaire assessing meniscal tear-related quality of life across three domains: Physical Symptoms (10 items), Sports/Recreation/Work/Lifestyle (4 items), and Emotions (2 items). Each item is scored from 0 (no problem) to 5 (extreme problem), with total scores transformed to a 0-100 scale where 0 represents the best possible status and 100 represents the worst possible status. Higher scores indicate worse outcomes.
Change from Baseline in Active Knee Range of Motion at 12 Month | Baseline, weekly during the 8-week intervention, and at 2-, 6-, and 12-months post commencement of intervention.
  Participant-initiated knee flexion-extension range measured in degrees using standardized goniometry, recording movement from full extension to maximum voluntary flexion.
Change from Baseline in Passive Knee Range of Motion at 12 Month | Baseline, weekly during the 8-week intervention, and at 2-, 6-, and 12-months post commencement of intervention
  Researcher-assisted knee flexion-extension range measured in degrees using standardized goniometry, recording movement from full extension to maximum assisted flexion without participants' muscle activation
Change from Baseline in 60-Second Sit-to-Stand Test Score (Number of Repetitions) at 12 Months | Baseline, weekly during the 8-week intervention, and at 2-, 6-, and 12-months post commencement of intervention.
  Quantifies lower limb functional strength and endurance by counting the maximum number of full sit-to-stand cycles completed in 60 seconds from a standardized-height chair. Higher counts indicate better functional performance.
Change from Baseline in 30-Second Step-Up Test Score (Number of Repetitions) at 12 Months | Baseline, weekly during the 8-week intervention, and at 2-, 6-, and 12-months post intervention
  The maximum number of complete step-up cycles performed in 30 seconds on a standardized step. Higher counts indicate better unilateral strength.
Change from Baseline in 30-Second Step-Down Test Score (Number of Repetitions) at 12 Months | Baseline, weekly during the 8-week intervention, and at 2-, 6-, and 12-months post commencement of intervention
  Quantifies unilateral lower limb strength by counting the maximum number of complete step-down cycles performed in 30 seconds on a standardized step. Higher counts indicate better unilateral strength and eccentric control.
Change from Baseline in Tissue Oxygenation 8 Weeks Using Photoacoustic Ultrasound Imaging | Weekly during the 8-week intervention
  Oxygenation saturation levels (%) measured by photoacoustic ultrasound around the meniscal tissue area.
Change from Baseline Vascularity Levels at 8 weeks using Photoacoustic Ultrasound Imaging. | Weekly during the 8-week intervention
  Vascularity levels (AU) measured by photoacoustic ultrasound around the meniscal tissue area.
Change from baseline skin temperature around the knee joint at 8 weeks using infrared thermography imaging. | Weekly during the 8-week intervention
Change from Baseline in Meniscal Morphology at 8 Weeks Using Ultrasound Imaging | Baseline and weekly during the 8-week intervention
  Meniscal structural integrity assessed via standardized ultrasound protocol using a validated 4-point scale where higher grades indicate worse pathology.
Number of participants with re-injury and associated ligament injuries, as assessed via both clinical examination and MRI. | Baseline to 6 months post commencement of intervention
  A re-injury or new ligament injury will be confirmed if both clinical examination indicates instability or significant changes from baseline, and MRI shows new or worsened structural damage compared to baseline images. We will document all instances of re-injury or new ligament injuries, including their nature and severity. The incidence of re-injuries and new ligament injuries will be compared between the PEMF and control groups, and we will analyze any correlation between meniscal healing status and the occurrence of re-injuries.
Change in Static Postural Control Assessed by Zebris Stance Analysis | Baseline, weekly during the 8-week intervention, and at 2-, 6-, and 12-months post intervention
  Quantitative postural control assessment during 10-second standing on the Zebris stance analysis system, which consists of a capacitance-based foot pressure platform inserted within a treadmill. Parameters include postural sway and weight distribution such as sway area, forefoot vs heel force ratio, left vs right symmetry
Change in Gait Function Assessed by Zebris Gait Analysis | Baseline, weekly during the 8-week intervention, and at 2-, 6-, and 12-months post intervention
  Quantitative gait analysis during 5-minute walking on the Zebris gait analysis system, which consists of a capacitance-based foot pressure platform inserted within a treadmill. Spatiotemporal parameters (gait speed, step length, stride length, cadence), dynamic balance (centre of pressure path length, lateral symmetry index), and load distribution metrics (peak heel/forefoot pressure, weight transfer timing) will be collected.
Change in Running Function Assessed by Zebris Gait Analysis | Baseline, weekly during the 8-week intervention, and at 2-, 6-, and 12-months post intervention
  Quantitative gait analysis during a 5-minute run on the Zebris gait analysis system, which consists of a capacitance-based foot pressure platform inserted within a treadmill. Spatiotemporal parameters (gait speed, step length, stride length, cadence), dynamic balance (centre of pressure path length, lateral symmetry index), and load distribution metrics (peak heel/forefoot pressure, weight transfer timing) will be collected.

CONTACTS AND LOCATIONS:
Locations (1):
- Room 124007, 10/F, Lui Chi Woo Clinical Sciences Building, Prince of Wales Hospital, Shatin, New Territories, Hong Kong SAR, China, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting 6 months after publication